CLINICAL TRIAL: NCT03306979
Title: Efficacy and Safety of N-acetylcysteine (NAC) in Patients With Mild Vascular Cognitive Impairment
Brief Title: Memory and Antioxidants in Vascular Impairment Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 241-2017
Record Dates: First submitted 2017-08-31; First posted 2017-10-11 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-03

CONDITIONS: Vascular Cognitive Impairment no Dementia
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Active Comparator): Participants randomized into the N-acetylcysteine arm will be receiving N-acetylcysteine for 24 weeks.
  Interventions: Drug: N Acetylcysteine
- Placebo (Placebo Comparator): Participants randomized into the placebo arm will be receiving placebo for 24 weeks.
  Interventions: Other: Placebo oral capsule

INTERVENTIONS:
Drug: N Acetylcysteine — Patients will be randomized to receive N Acetylcysteine (NAC) (four 600 mg capsules given as 2 capsules in the morning and 2 capsules in the evening). The initial NAC dosage will be 600mg/day (one 600mg capsule in the morning) for the first week, followed by 1,200 mg/day (one 600 mg capsule in the morning, one 600mg capsule in the evening) for the second week, followed by 1,800 mg/day (two 600mg capsules in the morning, one 600mg capsule in the evening) for third week, followed by 2,400mg/day (two 600mg capsules in the morning, two 600mg capsules in the evening) for the following 21 weeks.
  Other Names: NPN 80004844
  Arms: N-acetylcysteine
Other: Placebo oral capsule — Patients will receive four placebo capsules (lactose-based filler) given as 2 capsules in the morning and 2 capsules in the evening, which will be prepared to mimic the weight of the experimental capsules.The initial placebo dosage will be 600mg/day (one 600mg capsule in the morning) for the first week, followed by 1,200 mg/day (one 600 mg capsule in the morning, one 600mg capsule in the evening) for the second week, followed by 1,800 mg/day (two 600mg capsules in the morning, one 600mg capsule in the evening) for third week, followed by 2,400mg/day (two 600mg capsules in the morning, two 600mg capsules in the evening) for the following 21 weeks.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a 24-week randomized, double-blind, placebo-controlled parallel group design study involving Vascular cognitive impairment-no dementia (VCIND) patients to evaluate the efficacy and safety of oral NAC supplementation (2,400 mg daily) as an add-on therapy to improve cognitive function in patients undergoing cardiac rehabilitation (CR). The CR program consists of a harmonized aerobic and resistance training in a supervised group setting. Eligible patients will be randomized to receive NAC (four 600 mg capsules given as 2 capsules in the morning and 2 capsules in the evening) or matching placebo capsules. The initial NAC dosage will be 600mg/day (one 600mg capsule in the morning) for the first week, followed by 1,200 mg/day (one 600 mg capsule in the morning, one 600mg capsule in the evening) for the second week, followed by 1,800 mg/day (two 600mg capsules in the morning, one 600mg capsule in the evening) for third week, followed by 2,400mg/day (two 600mg capsules in the morning, two 600mg capsules in the evening) for the following 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 55-80 years.
* MoCA score of less than 28.
* Modest deficits (1 SD below population norm) in executive function, memory, processing speed, or working memory based on the 60-minute battery recommended by the NINDS-CSN.
* Speaks and understands English.
* Enrollment in the Cardiac Rehabilitation program at the University Health Network Toronto Rehabilitation Institute.

Exclusion Criteria:

* A history of stroke
* A history of epilepsy
* Uncontrolled asthma (requiring hospitalization or ER visit in the last 3 months by patient report)
* Uncontrolled diabetes (clinical determination)
* Severe hypo/hypertension (clinical determination)
* Uncontrolled hypercholesterolemia (clinical determination)
* Presence of significant medical illnesses (Severely disturbed liver function, Severely disturbed kidney function, Severely disturbed lung function, HIV, HBV and/or HCV infection, Malignant tumors)
* A current neurological condition (Parkinson's disease, Multiple sclerosis, Significant traumatic brain injury)
* Major psychiatric condition (Current major depressive disorder, Schizophrenia, Bipolar disorder, Substance use disorder (alcohol abuse, heavy smoking (20 cigarettes or more/day))
* Contraindication to MRI or MRS (e.g. metal in body, pacemaker).
* Contraindication to NAC (documented allergy) or allergy to lactose.
* Daily Nitroglycerin use.
* Bleeding disorders (e.g. hemophilia, Thrombotic Thrombocytopenic Purpura) and/or elective surgery within 30 days.
* Volunteers who currently participate in another pharmacological study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krista L Lanctôt, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-acetylcysteine | Placebo
Started (A participant was randomized however dropped out prior to actually starting any study drug so is not included in this count.) | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.0) | 68.0 (7.5) | 67.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 17 | 24 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Arab/Middle Eastern | 2 | 0 | 2
  Ethnicity: Asian/South Asian | 5 | 7 | 12
  Ethnicity: Black/African American | 3 | 1 | 4
  Ethnicity: Caucasian/European | 19 | 21 | 40
  Ethnicity: Other (mixed) | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 29 | 30 | 59
Executive Function [Mean (Standard Deviation); unit: z-score] — A composite score that included tests of verbal (phonemic) fluency, category (semantic) fluency, and the trail making test B.
  A Z-score was computed based on published age-matched norms, and a composite Z-score was calculated. A Z-score of 0 represents the population mean, with higher Z-score representing better cognitive function.
  z-score | -0.54 (0.68) | -0.48 (0.48) | -0.52 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Change in Executive Function
Description: Differences in executive function composite z scores between experimental and placebo groups at 6 months. Executive function will be based on the trail test B, phonemic fluency, and semantic fluency found in the 60-minute battery recommended by the National Institute of Neurological Disorders and Stroke-Canadian Stroke Network (NINDS-CSN) harmonized standards. A Z-score was computed based on published age-matched norms, and a composite Z-score was calculated. Higher z score represents better cognitive function.
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 29 | 30
z-score | 0.32 [0.20 to 0.52] | 0.36 [0.20 to 0.52]

2. Secondary Outcome: Change in Processing Speed
Description: Differences in processing speed composite z scores between experimental and placebo groups at 6 months. Processing speed will be based on the symbol digit modalities test found in the 60-minute battery recommended by the National Institute of Neurological Disorders and Stroke-Canadian Stroke Network (NINDS-CSN) harmonized standards. A z-score was computed based on published age-matched norms. Higher z-score represents better cognitive function.
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 29 | 30
Z-score | 0.03 [-0.16 to 0.35] | 0.17 [-0.02 to 0.35]

3. Secondary Outcome: Change in Memory
Description: Differences in memory composite z scores between experimental and placebo groups at 6 months. Memory will be based on the Hopkins Verbal Learning Test found in the 60-minute battery recommended by the National Institute of Neurological Disorders and Stroke-Canadian Stroke Network (NINDS-CSN) harmonized standards. A z-score was computed based on published age-matched norms. Higher z-scores represent better cognitive function.
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 29 | 30
z-score | 0.03 [-0.21 to 0.27] | -0.10 [-0.21 to 0.19]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | N-acetylcysteine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 21/29 | 20/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine (N=29) | Placebo (N=30)
Dyspepsia (Gastrointestinal disorders) | 10 | 6
Diarrhea (Gastrointestinal disorders) | 2 | 5
Headache (General disorders) | 8 | 5
Epigastric discomfort (Gastrointestinal disorders) | 9 | 7
Nausea (General disorders) | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Tinnitus (Ear and labyrinth disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03306979/Prot_SAP_000.pdf